CLINICAL TRIAL: NCT05916222
Title: The Effects of Caregiver Training on Dynamic Temporal and Tactile Cueing (DTTC) Treatment Outcomes in Childhood Apraxia of Speech (CAS)
Brief Title: The Effects of Caregiver Training on DTTC Treatment Outcomes in CAS
Acronym: DTTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: Hofstra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A22-0040-001
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Childhood Apraxia of Speech
Keywords: Children; Speech; Intervention
MeSH Terms: conditions — Apraxias; Speech

STUDY DESIGN:
Intervention Model Description: This proposed work is multisite parallel-group randomized control trial (RCT) that aims to investigate the impact of parent/caregiver involvement on DTTC treatment outcomes in children with CAS. Participants will be seen in two groups: 1) Direct Training Group (DTTC + Home Practice + Direct Caregiver Training); 2) Indirect Training Group (DTTC + Home Practice + Indirect Caregiver Training).
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessors will be unaware of participant grouping (i.e., Direct Training Group, Indirect Training Group), treatment phase (i.e., baseline, treatment, follow-up), or status of words (i.e., treated, generalization words).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Training (DTTC + Home Practice) (Active Comparator): Children in the Indirect Training Arm will receive DTTC treatment 2x/week administered by an SLP for 8 weeks. Parent/caregivers in this Arm will complete an online, self-paced educational module on CAS prior to the start of treatment, observe all treatment sessions, and review home practice guidelines with the clinician at the end of each therapy session. Parent/caregivers will engage their children in home practice during the treatment phase and follow-up phase. Home practice will consist of 30-minute practice sessions 3x/week during the 8-week treatment phase and 6x/week during the 4-week follow-up phase.
  Interventions: Behavioral: Dynamic Temporal and Tactile Cueing (DTTC)
- Direct Training (DTTC + Coaching + Home Practice) (Experimental): Children in the Direct Training Arm will receive DTTC treatment 2x/week for 8 weeks with half of each session administered only by the SLP. In the other half of the session, DTTC will be administered by the parent/caregiver with online coaching by the SLP. During the coaching portion of treatment sessions, the SLP will provide direct training to guide the parent/caregiver in the administration of DTTC to support home practice sessions. Parent/caregivers in this Arm will also complete an online, self-paced educational module on CAS prior to the start of treatment and review home practice guidelines with the clinician at the end of each therapy session. Parent/caregivers will engage their children in home practice during the treatment phase and follow-up phase. Home practice will consist of 30-minute practice sessions 3x/week during the 8-week treatment phase and 6x/week during the 4-week follow-up phase.
  Interventions: Behavioral: Dynamic Temporal and Tactile Cueing (DTTC)

INTERVENTIONS:
Behavioral: Dynamic Temporal and Tactile Cueing (DTTC) — DTTC is a motor-based intervention where the client watches, listens to and imitates the clinician (Strand, 2020). Treatment follows a temporal hierarchy where children receive multisensory cueing to establish accurate movements. First, the child imitates the clinician's production. If inaccurate, the child simultaneously produces the target with the clinician while cueing is provided. Upon achieving accuracy within simultaneous productions, the target is practiced within direct imitation while the clinician adds/fades cues based on the child's productions. When the child accurately produces the target in direct imitation, the target is practiced with varied prosody. Next, the target is practiced within delayed imitation where a child produces a word following a 2-3 second delay after the clinician's production. Upon accurately producing the target at all levels, the word is practiced within spontaneous productions.
  Other Names: DTTC

SUMMARY:
The goal of this clinical trial is to investigate the impact of direct vs. indirect caregiver training on treatment outcomes following a period of Dynamic Temporal and Tactile Cueing (DTTC) intervention combined with home practice in childhood apraxia of speech (CAS). Forty children with CAS, between the ages of 2;5 and 7;11 years of age, will be recruited for this study. All children will receive DTTC treatment at the frequency of standard care (2x/week) in a university clinic over and 8-week period. Participants will be randomly assigned to one of two groups: the Direct Training Group; the Indirect Training Group. All caregivers will complete an educational module about CAS, will observe all sessions, and will engage in home practice with their children. Caregivers in the Direct Group will receive coaching in the use of DTTC with their child during a portion of each treatment session to support home practice, whereas those in the Indirect Group will not receive detailed guidance for home practice. Caregivers in both groups will practice at home with their children during the treatment phase (3x/week). Following the treatment phase, home practice will continue at a higher frequency (6x/week) during a 4-week follow-up phase. Treatment outcomes will be compared between groups.

DETAILED DESCRIPTION:
Forty children with CAS, between 2;5 and 7;11 years of age will receive DTTC treatment 2x/week over an 8-week period along with home practice with a caregiver. Prior to treatment, all caregivers will complete an online self-guided educational module about CAS and DTTC. Participants will be randomized to one of two groups: 1) Direct Training Group (DTTC + Home Practice + Direct Caregiver Training); 2) Indirect Training Group (DTTC + Home Practice + Indirect Caregiver Training).

Children in the Direct Training Group will receive DTTC treatment during one half of each session administered only by the SLP, while the caregiver observes. DTTC will be administered by the caregiver with direct coaching by the speech language pathologist (SLP) in the other half of the session. Children in the Indirect Training Group will only receive DTTC treatment administered by the SLP, while the caregiver observes. In both groups, caregivers will review home practice guidelines with the clinician at the end of each therapy session, and engage in home practice with their children. Home practice will consist of 30-minute practice sessions 3x/week during the 8-week treatment phase and 6x/week during the 4-week follow-up phase. Caregivers in the Direct Training Group will be provided specific guidance regarding practice techniques, whereas caregivers in the Indirect Training Group will only be provided treatment words to be practiced at home and instructed to apply what they have observed during SLP-administered DTTC.

Probe data will be collected during the Pre-Treatment, Treatment and Follow-Up phases. The study duration is 16 weeks in total duration, for all participants. Probe words will consist of 20 potential treated items to evaluate treatment gains and 30 generalization items to assess carryover of treatment gains to untreated words.

The study will address the following aims:

Aim 1: Quantify the effects of direct vs. indirect caregiver training during a period of DTTC combined with home practice on whole word accuracy in treated and generalization probes at post-treatment and maintenance.

Aim 2: Quantify the effects of direct vs. indirect caregiver training during a period of DTTC combined with home practice on phoneme accuracy in treated words and generalization probes at post-treatment and maintenance.

Aim 3: Quantify the effects of direct vs. indirect caregiver training during a period of DTTC combined with home practice on speech intelligibility at post-treatment and maintenance.

Aim 4: Quantify the effects of direct vs. indirect caregiver training during a period of DTTC combined with home practice on functional communication at post-treatment and maintenance.

ELIGIBILITY:
Child Eligibility

Inclusion Criteria

1. 2;6-7;11 years of age at the start of treatment
2. English as the primary and preferred language
3. Primary speech diagnosis of CAS based on auditory-perceptual, expert diagnosis and/or Dynamic Evaluation of Motor Speech Skills (DEMSS) score classification of "significant evidence of CAS" with score <323

Exclusion Criteria

1. Concomitant disorders including autism spectrum disorder, global development delay, or intellectual disability, Down syndrome, or other genetic condition (diagnosis of Attention Deficit and Hyperactivity Disorder (ADHD) is allowable if the child can attend in sessions with medication and/or strategies)
2. Primary diagnosis of dysarthria or other speech sound disorder (e.g., phonological impairment).
3. Oral structural anomalies
4. Hearing impairment
5. Uncorrected visual impairment
6. Receiving speech treatment elsewhere during the period of the study. Language or Augmentative and Alternative Communication (AAC) treatment is permitted.
7. Receptive Language Index standard score less than 70 on the Receptive-Expressive Emergent Language Test - 4th Edition (REEL-4), Clinical Evaluation of Language Fundamentals - Preschool 3rd Edition (CELF-P3), or Clinical Evaluation of Language Fundamentals - 5th Edition (CELF-5), as appropriate for participant's age.
8. Cognitive standard score less than 70 on the Developmental Assessment of Young Children (DAYC) - ages 2;0 - 5;11, Nonverbal Index of Reynolds Intellectual Assessment Scales - 2nd Edition - age 6;0 - 7;11

Ages: 24 Months to 95 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in word accuracy | Pre- to post-treatment (16 treatment sessions over 8 weeks); 1-week and 4-week post-treatment follow-up
  A multi-factor whole-word accuracy measure (Multilevel word Accuracy Composite Scale (MACS); Case et al., in press) of segmental accuracy, word shape maintenance, prosodic accuracy, and smoothness/fluency of movement transitions will be calculated for treated and generalization words. A MACS score ranges from 0 (all inaccurate) to 1.0 (all accurate). The higher the MACS score is to 1, the more accurate the production would be for that word. Judgments of word accuracy will be made by anonymous raters. The MACS will be used to address Aim 1(effect of DTTC combined with parent/caregiver coaching on speech production accuracy).

SECONDARY OUTCOMES:
Changes in phoneme accuracy | Pre- to post-treatment (16 treatment sessions over 8 weeks); 1-week and 4-week post-treatment follow-up
  Percentage of accurate phonemes will be calculated for treated and generalization words. Judgments of phoneme accuracy will be made by anonymous raters. Phoneme accuracy will be used to address Aim 2 (effect of DTTC combined with parent/caregiver coaching on phoneme accuracy).
Changes in speech intelligibility | Pre- to post-treatment (16 treatment sessions over 8 weeks); 1-week and 4-week post-treatment follow-up
  The Intelligibility in Context Scale (ICS; McLeod et al., 2012), a parent report measure of children's intelligibility, will be administered. An ICS score ranges from 1.0 (low intelligibility) to 5.0 (high intelligibility).The ICS will be used to address Aim 3 (effect of DTTC combined with parent/caregiver coaching on speech intelligibility).
Changes in the FOCUS-34 score | Pre- to post-treatment (16 treatment sessions over 8 weeks); 1-week and 4-week post-treatment follow-up
  The Functional Outcomes on Communication Under Six (FOCUS-34; Thomas-Stonell et al., 2015), a parent survey measure, will be administered to examine change in children's communication skills. The FOCUS-34 will be used to address Aim 4 (effect of DTTC combined with parent/caregiver coaching on functional communication).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hofstra University, Hempstead, New York
  - New York University, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data tied to the primary and secondary outcome measures will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months following publication. No end date.
Access Criteria: Researchers and speech language pathologists who provide a methodologically sound proposal. Proposals should be directed to maria.grigos@nyu.edu and julie.case@hofstra.edu. To gain access, data requestors will need to complete and sign a data sharing agreement.

REFERENCES:
- [Background] Strand EA. Dynamic Temporal and Tactile Cueing: A Treatment Strategy for Childhood Apraxia of Speech. Am J Speech Lang Pathol. 2020 Feb 7;29(1):30-48. doi: 10.1044/2019_AJSLP-19-0005. Epub 2019 Dec 17. PMID 31846588
- [Background] Case J, Wang EW, Grigos MI. The Multilevel Word Accuracy Composite Scale: A Novel Measure of Speech Production in Childhood Apraxia of Speech. Am J Speech Lang Pathol. 2023 Aug 17;32(4S):1866-1883. doi: 10.1044/2023_AJSLP-22-00166. Epub 2023 May 17. PMID 37195724
- [Background] McLeod S, Harrison LJ, McCormack J. The intelligibility in Context Scale: validity and reliability of a subjective rating measure. J Speech Lang Hear Res. 2012 Apr;55(2):648-56. doi: 10.1044/1092-4388(2011/10-0130). Epub 2012 Jan 3. PMID 22215036
- [Background] Thomas-Stonell N, Washington K, Oddson B, Robertson B, Rosenbaum P. Measuring communicative participation using the FOCUS(c): Focus on the Outcomes of Communication Under Six. Child Care Health Dev. 2013 Jul;39(4):474-80. doi: 10.1111/cch.12049. PMID 23763248